CLINICAL TRIAL: NCT01554800
Title: An Intravenous, Open-label, Single-dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of rhLCAT in Subjects With Coronary Artery Disease
Brief Title: Effect of ACP-501 on Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Subjects With Coronary Artery Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP 501-01; 12-H-0092 (Other: NIH)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2013-01

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Lecithin Cholesterol Acyl Transferase; LCAT; rhLCAT; Enzyme replacement therapy; High-Density Lipoprotein (HDL); Cholesterol; Cholesterol ester; LCAT Deficiency
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Lecithin Cholesterol Acyltransferase Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACP-501 (Experimental)
  Interventions: Drug: ACP-501

INTERVENTIONS:
Drug: ACP-501 — A single dose infusion

SUMMARY:
This study is a phase 1, intravenous, open-label, single-dose escalation study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of ACP-501 (recombinant human Lecithin Cholesterol Acyl Transferase (rhLCAT)) in subjects with coronary artery disease (CAD). Four cohorts consisting of 4 subjects each will receive one dose of ACP-501. The dose will be escalated by cohort.

DETAILED DESCRIPTION:
After signing informed consent, subjects entered into the trial will be followed for up to 8 weeks which includes: up to 4 weeks screening, entry criteria assessments on Day 0 and single-dose IV infusion on Day 1, and 4 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* A history of stable documented CAD
* Currently non-smoking males and females ages 30 to 85 years inclusive.

  o Female subjects of child-bearing potential (neither pregnant nor breast-feeding) must be using adequate birth control during study conduct.
* Chronic concomitant medications must be stable for at least 2 months prior to screening
* HDL-C < 50 mg/dL for men and < 55 mg/dL for women
* Body Mass Index (BMI) of approximately 18 to 35 kg/m^2; and a total body weight >= 50 kg (110 lbs) and <= 110 kg (approximately 242 lbs)

Exclusion Criteria:

* Myocardial infarction, stroke, or coronary intervention/revascularization procedure within 6 months prior to dosing.
* Chronic heart failure (> New York Heart Association (NYHA) Functional Classification II).
* Ventricular tachyarrhythmias.
* Uncontrolled Type 2 (HbA1c > 8.5%) or Type 1 diabetes mellitus.
* History of febrile illness within 5 days prior to dosing.
* History of regular alcohol consumption exceeding 10 drinks per week.
* 12-lead ECG demonstrating QTc > 500 msec at screening.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Summary of Participants Experience with Safety and Tolerability | Day 1 to Day 28
  Safety and tolerability of a single dose of ACP-501 as determined by adverse event reporting, clinical laboratory results, vital signs, physical examination, and electrocardiograms (ECGs).

SECONDARY OUTCOMES:
Pharmacokinetic profile | Hours 0, 1, 6, 12, 24, 48, 72, 96, 168
Change in High-Density Lipoprotein-Cholesterol (HDL-C) value following a single dose | Hours 0, 1, 6, 12, 24, 48, 72, 96, 168

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular and Pulmonary Branch (CPB) of NIH, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Shamburek RD, Bakker-Arkema R, Shamburek AM, Freeman LA, Amar MJ, Auerbach B, Krause BR, Homan R, Adelman SJ, Collins HL, Sampson M, Wolska A, Remaley AT. Safety and Tolerability of ACP-501, a Recombinant Human Lecithin:Cholesterol Acyltransferase, in a Phase 1 Single-Dose Escalation Study. Circ Res. 2016 Jan 8;118(1):73-82. doi: 10.1161/CIRCRESAHA.115.306223. Epub 2015 Dec 1. PMID 26628614